CLINICAL TRIAL: NCT01919580
Title: Observational Study on the Carcinogenesis of Gα12 in Oral Cancer, and Chemopreventive Possibility for the Treatment of Oral Cancer Using Ga12 Inhibitor.
Brief Title: Study on the Carcinogenesis of Gα12 in Oral Cancer, and the Treatment of Oral Cancer Using Ga12 Inhibitor.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112057RIB
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Carcinogenesis; Oral Cancer
Keywords: Gα12; Oral cancer
MeSH Terms: conditions — Carcinogenesis; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — tissue, serum, saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal team: Subjects who have problem at third molar of impacted tooth need to receive a surgery with general anesthesia.
  Subjects must:
  Should have a blood exam (20ml) before the surgery.
  Site staff must:
  Collect subjects' saliva once a day (in the morning before breakfast) for 3 consecutive days.
  Collect a 0.5x0.5Cm2 tissue sample around third molar during the surgery.
- Oral dysplasia: Subjects who are diagnosed with dysplasia of oral cavity.
  Subjects must:
  Should have a blood exam (20ml/each time) before the surgery and 3 months after the surgery.
  In the case the disease recurs after the surgery, subjects need to receive the surgery again and take another blood exam before the surgery and 3 months after the surgery.
  Before the surgery site staff must:
  Collect subjects' saliva once a day (in the morning before breakfast) for 3 consecutive days.
  Collect a 0.5x0.5Cm2 tissue sample of the tumor during the surgery.
- Oral cancer: Subjects who suffer from oral cancer.
  Subjects must:
  Should have a blood exam (20ml/each time) before the surgery and 3 months after the surgery.
  In the case the disease recurs after the surgery, subjects need to receive the surgery again and take another blood exam before the surgery and 3 months after the surgery.
  Before the surgery site staff must:
  Collect subjects' saliva once a day (in the morning before breakfast) for 3 consecutive days.
  Collect a 0.5x0.5Cm2 tissue sample of the tumor during the surgery.

SUMMARY:
Study on the carcinogenesis of Gα12 in oral cancer, and chemopreventive possibility for the treatment of oral cancer using Ga12 inhibitor.

DETAILED DESCRIPTION:
To find out if there is prognostic value which to the performance of Gα12 of oral cancer in Taiwan and provide some reference for future treatment.

We anticipate to enroll 40 persons with normal oral mucosa, 65 persons with oral dysplasia and 150 persons with oral cancer and collect the tissue which was stained for pathological sections over a 3 year period.

We also collect the blood and saliva samples from patients and the results along with patient-specific information such as tumor phases, tumor size, lymph node metastasis, cancer metastasis, prognosis and betel nut chewing, smoking and drinking habits and other parameters are statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Dysplasia or cancer of the oral cavity.

Exclusion Criteria:

* pregnant woman

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical center
Sampling Method: Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Carcinogenesis of Gα12 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Jung Cheng, DDS, MS, PhD, Principal Investigator
Locations (1):
- National Taiwan University Hospital research Ethics Committee, Taipei, Taiwan

REFERENCES:
- [Background] Dolezalova H, Shankar G, Huang MC, Bikle DD, Goetzl EJ. Biochemical regulation of breast cancer cell expression of S1P2 (Edg-5) and S1P3 (Edg-3) G protein-coupled receptors for sphingosine 1-phosphate. J Cell Biochem. 2003 Mar 1;88(4):732-43. doi: 10.1002/jcb.10394. PMID 12577307
- [Background] Dorsam RT, Gutkind JS. G-protein-coupled receptors and cancer. Nat Rev Cancer. 2007 Feb;7(2):79-94. doi: 10.1038/nrc2069. PMID 17251915
- [Background] Etienne-Manneville S, Hall A. Rho GTPases in cell biology. Nature. 2002 Dec 12;420(6916):629-35. doi: 10.1038/nature01148. PMID 12478284
- [Background] Friedl P, Wolf K. Tumour-cell invasion and migration: diversity and escape mechanisms. Nat Rev Cancer. 2003 May;3(5):362-74. doi: 10.1038/nrc1075. PMID 12724734
- [Background] Gilman AG. G proteins: transducers of receptor-generated signals. Annu Rev Biochem. 1987;56:615-49. doi: 10.1146/annurev.bi.56.070187.003151. No abstract available. PMID 3113327
- [Background] Gohla A, Offermanns S, Wilkie TM, Schultz G. Differential involvement of Galpha12 and Galpha13 in receptor-mediated stress fiber formation. J Biol Chem. 1999 Jun 18;274(25):17901-7. doi: 10.1074/jbc.274.25.17901. PMID 10364236
- [Background] Gu JL, Muller S, Mancino V, Offermanns S, Simon MI. Interaction of G alpha(12) with G alpha(13) and G alpha(q) signaling pathways. Proc Natl Acad Sci U S A. 2002 Jul 9;99(14):9352-7. doi: 10.1073/pnas.102291599. Epub 2002 Jun 20. PMID 12077299
- [Background] Meigs TE, Fedor-Chaiken M, Kaplan DD, Brackenbury R, Casey PJ. Galpha12 and Galpha13 negatively regulate the adhesive functions of cadherin. J Biol Chem. 2002 Jul 5;277(27):24594-600. doi: 10.1074/jbc.M201984200. Epub 2002 Apr 25. PMID 11976333
- [Background] Moers A, Nurnberg A, Goebbels S, Wettschureck N, Offermanns S. Galpha12/Galpha13 deficiency causes localized overmigration of neurons in the developing cerebral and cerebellar cortices. Mol Cell Biol. 2008 Mar;28(5):1480-8. doi: 10.1128/MCB.00651-07. Epub 2007 Dec 17. PMID 18086886
- [Background] Parks S, Wieschaus E. The Drosophila gastrulation gene concertina encodes a G alpha-like protein. Cell. 1991 Jan 25;64(2):447-58. doi: 10.1016/0092-8674(91)90652-f. PMID 1899050
- [Background] Radeff-Huang J, Seasholtz TM, Matteo RG, Brown JH. G protein mediated signaling pathways in lysophospholipid induced cell proliferation and survival. J Cell Biochem. 2004 Aug 1;92(5):949-66. doi: 10.1002/jcb.20094. PMID 15258918
- [Background] Radhika V, Hee Ha J, Jayaraman M, Tsim ST, Dhanasekaran N. Mitogenic signaling by lysophosphatidic acid (LPA) involves Galpha12. Oncogene. 2005 Jun 30;24(28):4597-603. doi: 10.1038/sj.onc.1208665. PMID 15856019
- [Background] Xu J, Wang F, Van Keymeulen A, Herzmark P, Straight A, Kelly K, Takuwa Y, Sugimoto N, Mitchison T, Bourne HR. Divergent signals and cytoskeletal assemblies regulate self-organizing polarity in neutrophils. Cell. 2003 Jul 25;114(2):201-14. doi: 10.1016/s0092-8674(03)00555-5. PMID 12887922
- [Background] Yu YP, Landsittel D, Jing L, Nelson J, Ren B, Liu L, McDonald C, Thomas R, Dhir R, Finkelstein S, Michalopoulos G, Becich M, Luo JH. Gene expression alterations in prostate cancer predicting tumor aggression and preceding development of malignancy. J Clin Oncol. 2004 Jul 15;22(14):2790-9. doi: 10.1200/JCO.2004.05.158. PMID 15254046
- [Result] Buhl AM, Johnson NL, Dhanasekaran N, Johnson GL. G alpha 12 and G alpha 13 stimulate Rho-dependent stress fiber formation and focal adhesion assembly. J Biol Chem. 1995 Oct 20;270(42):24631-4. doi: 10.1074/jbc.270.42.24631. PMID 7559569
- [Result] Chan AM, Fleming TP, McGovern ES, Chedid M, Miki T, Aaronson SA. Expression cDNA cloning of a transforming gene encoding the wild-type G alpha 12 gene product. Mol Cell Biol. 1993 Feb;13(2):762-8. doi: 10.1128/mcb.13.2.762-768.1993. PMID 8423800